CLINICAL TRIAL: NCT02851238
Title: Driving Pressure Limited Ventilation Decreases Postoperative Pulmonary Complications in One-Lung Ventilation: Randomized Controlled Study
Brief Title: Driving Pressure and Postoperative Pulmonary Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Joo Ahn, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SMC 2016-05-107-003
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: One-Lung Ventilation; Postoperative Respiratory Complications; Driving Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Protective Ventilation (No Intervention): The control arm receives existing conventional protective ventilation with tidal volume of 6mL/kg of ideal body weight and positive end expiratory ventilation of 5cmH2O during one-lung ventilation
- Driving Pressure Limited Ventilation (Experimental): The intervention arm receives driving pressure limited ventilation during one-lung ventilation
  Interventions: Other: Driving Pressure Limited Ventilation

INTERVENTIONS:
Other: Driving Pressure Limited Ventilation — Positive end expiratory pressure is adjusted to minimize driving pressure, plateau pressure minus end expiratory pressure from 2 to 10 cmH2O during one-lung ventilation
  Arms: Driving Pressure Limited Ventilation

SUMMARY:
This study aims to prove that driving pressure limited ventilation is superior in preventing postoperative pulmonary complications to existing protective ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 19 years
* Patient who undergoes one-lung ventilation for thoracic surgery

Exclusion Criteria:

* The American Society of Anesthesiologists (ASA) Physical Status classification greater than or equal to 4
* Patient who is contraindicated with application of positive end expiratory pressure
* Patient who rejects being enrolled in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative pulmonary complications | within the first 3 days after surgery
  Patient is regarded to have postoperative pulmonary complication when 4 or more positive variables exists according to Melbourne Group Scale.

SECONDARY OUTCOMES:
Partial pressure of oxygen in arterial blood | during surgery
The ratio of partial pressure arterial oxygen and fraction of inspired oxygen | on the first postoperative day
  The ratio will be obtained from the first arterial blood gas analysis on the first postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Ahn, Ph.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea